CLINICAL TRIAL: NCT00926068
Title: Safety and Efficacy of HO/03/03 10μg in the Treatment of Plantar Neuropathic Diabetic Foot Ulcers (Truheal)
Brief Title: Safety and Efficacy of HO/03/03 10μg in the Treatment of Plantar Neuropathic Diabetic Foot Ulcers
Acronym: Truheal
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: HealOr (Industry)
Collaborators: Clinigene International Ltd (Industry); Cato Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HO-09-01
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes Mellitus; Foot Ulcer; DFU; Wound healing
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HO/03/03 10µg (Experimental)
  Interventions: Drug: HO/03/03 10µg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HO/03/03 10µg
  Arms: HO/03/03 10µg
Drug: Placebo
  Arms: Placebo

SUMMARY:
A prospective, double blind, randomized, placebo controlled, outpatient, parallel group comparison trial to assess the safety and efficacy of HO/03/03 10µg versus Placebo, applied topically once daily for up to 14 weeks in at least 196 subjects diagnosed with Diabetes Mellitus and having a single target non-healing Plantar Neuropathic Diabetic Foot Ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years, extremes included
2. Diagnosed with Diabetes Mellitus Type 1 or Type 2
3. Having a documented single target non-healing Plantar Neuropathic Diabetic Foot Ulcer with a minimal duration of 4 weeks prior to the informed consent signature
4. Ulcer size at randomization:

   * Wagner grade 1, between 2.0 cm2 to 10 cm2, extremes included or;
   * Wagner grade 2, between 1.0 cm2 to 10 cm2, extremes included;
5. Single target, ulcer on the study foot:

   * Wagner grade 1 or;
   * Wagner grade 2 (does not involve abscess or osteomyelitis);
6. Target ulcer area decreased by ≤ 30% OR ≤ 0.1 cm/wk edge healing rate measured after debridement at screening to after debridement if clinically indicated at randomization.
7. Glycosylated Haemoglobin A1c (HbA1c) ≤ 12%;
8. Ankle to Brachial Index (ABI) on study foot:

   * 0.7 ≤ ABI ≤ 1.2 or
   * ABI > 1.2 and toe pressure > 50 mm Hg (ABI measured by Doppler; toe blood pressure measured by toe cuff);
9. Diabetic Neuropathy is confirmed by neurological testing
10. Subject should be available for the entire study period, and be able and willing to adhere to protocol requirements
11. Subject has signed the informed consent form prior to any study protocol related procedure

Exclusion Criteria:

Subjects meeting one or more of the following criteria cannot be selected:

1. Anamnesis of current or recent past (within the last 2 years) abuse of alcohol, barbiturates, benzodiazepines, amphetamines, narcotics, cocaine, psychoactive drugs or other abused substances that will interfere with treatment compliance
2. Use of growth factors, skin graft or participation in an investigational study within the last 30 days prior to the beginning of the screening period
3. Females who are pregnant, lactating, of child-bearing potential, or post-menopausal for less than 2 years and not using a medically approved method of contraception or females who test positive on a blood-based pregnancy test
4. Have a documented medical history of HIV, HBV or HCV
5. Have a documented medical history of a significant cardiac, pulmonary, gastrointestinal, endocrine (other than Diabetes Mellitus type 1 or 2), metabolic, neurological, hepatic or nephrologic disease and/or receiving dialysis
6. Anaemia (Haemoglobin < 9 gram/dL for females or Haemoglobin < 10 gram/dL for males) or White Blood Cells count > 11,000/μL or Platelets count < 100,000/μL or impaired renal function (Creatinine > 3 mg/dL) or liver function tests > 3 times upper normal lab values or any indication of malnourishment (Albumin < 2.8 g/dL) or any other clinically significant biochemistry, haematology and urinalysis tests;
7. Had any clinically significant illness during the last 4 weeks prior to the screening period;
8. Have a current malignancy or a past malignancy in the last 5 years other than Basal Cell Carcinoma or is treated by radio/chemotherapy
9. Have any signs of clinical infection in the wound (which could be linked to raised body temperature, abscess, osteomyelitis, necrosis or erythema)
10. Had any antibiotic treatment during the screening period;
11. Had evidence of infection or osteomyelitis on a plain foot x-ray at screening;
12. Is bed-ridden or unable to come to the clinic;
13. Have more than one target non-healing Diabetic Foot Ulcer per subject;
14. Plantar Neuropathic DFU is located on an active Charcot foot;
15. Have hind foot ulcer or have a foot deformity/condition preventing the use of offload footwear;
16. Had a leg revascularization surgery within the last 6 months or be a candidate for revascularization surgery during the course of the study;
17. Glucocorticosteroid treatment (Prednisone >10 mg/day or its equivalent)
18. Inability to stop alternative wound healing treatment (e.g. Becaplermin or other topical products) following debridement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Complete ulcer closure | Up to 14 weeks inclusive
  Time to Event Analysis that determines time for incidence of 100% study wound closure per unit of time (days) and the incidence of 100% wound closure per unit of time using the log rank test.

SECONDARY OUTCOMES:
Percent change in wound area at 4 weeks | 4 weeks
75% wound closure by or on Study Week 14 | Up to 14 weeks inclusive
Incidence of adverse events, changes in vital signs, physical examination, electrocardiogram and laboratory tests from baseline to termination. | 14 weeks
Incidence of 100% Closure tested by the Fisher exact 2-tailed test | Up to 14 weeks inclusive
Percent change in granulation tissue at 4 weeks | 4 weeks
Incidence of improved ulcers

CONTACTS AND LOCATIONS:
Locations (33):
- United States (19):
  - Phoenix VA Healthcare System, Phoenix, Arizona
  - Center For Clinical Research, Castro Valley, California
  - Dr. Ian Gordon, Long Beach, California
  - Advanced Clinical Research, Los Angeles, California
  - Innovative Medical Technologies, LLC, Los Angeles, California
  - California School of Podiatric Medicine at Samuel Merritt University, Oakland, California
  - North American Centre for Limb Preservation, New Haven, Connecticut
  - Bay Pines VA Healthcare System-Wound Clinic Bay Pines VA Healthcare System-Research Pharmacy, Bay Pines, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Doctors Research Network, Miami, Florida
  - Capt. James A. Lovell Federal Health Care Center, North Chicago, Illinois
  - Deaconess Clinic Downtown-Research Institute, Evansville, Indiana
  - St. Vincent Wound Care Center IDI Research, Indianapolis, Indiana
  - Cambridge Hospital, Cambridge, Massachusetts
  - Center for Curative & Palliative Wound Care Calvary Hospital, New York, New York
  - Armstrong County Memorial Hospital Snyder Institute for Vascular Health and Research, Kittanning, Pennsylvania
  - Paddington Testing Company, Philadelphia, Pennsylvania
  - Martin Foot and Ankle, York, Pennsylvania
  - Complete Family Foot Care, McAllen, Texas
- India (14):
  - Medanta, Gurgaon, Haryana
  - Jain Institute of Vascular Sciences, Bangalore, Karnataka
  - Karnataka Institute of Diabetology, Bangalore, Karnataka
  - St.John's Hospital, Bangalore, Karnataka
  - Belgaum Diabetes Centre, Belagavi, Karnataka
  - Vinaya Hospital and Research Centre, Mangalore, Karnataka
  - Kunnamkulam Eye and Diabetes Centre, Thrissur, Kerala
  - OM Shree Swami Samarth Hospital, Pune, Maharashtra
  - Patil Hospital, Pune, Maharashtra
  - MV Hospital for Diabetes Pvt Ltd, Chennai, Tamil Nadu
  - Dr. V Seshiah Diabetes Research Institute, Chennai, Tamil Nadu
  - Christian Medical College, Vellore, Tamil Nadu
  - SK Diabetes Research & Education Center, Kolkata, West Bengal
  - Advanced Medicare & Research Institute, Kolkata